CLINICAL TRIAL: NCT04117334
Title: Determining the Best Indications for Initiating Brace Treatment for Adolescent Idiopathic Scoliosis
Brief Title: Determining Best Indications for Bracing for Adolescent Idiopathic Scoliosis
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: PB version 1.0
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Bracing; Cost-effectiveness; Adolescent idiopathic scoliosis
MeSH Terms: interventions — Braces

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bracing AIS patients: These are patients undergoing brace treatment for AIS
  Interventions: Other: Bracing

INTERVENTIONS:
Other: Bracing

SUMMARY:
This is a prospective study for Investigating the cost-effectiveness of current bracing protocols for adolescent idiopathic scoliosis (AIS). It is hypothesized that aggressive management of adolescent idiopathic scoliosis (AIS) including early bracing at mild curve magnitudes and surgery at 40 degrees is more cost-effective while maintaining similar health quality of life. Scoliosis Research Society 22-item and EuroQol- 5 dimension questionnaires and direct/indirect medical costs will be utilized for the cost-effectiveness analysis and health related quality of life assessment. The findings of this study have the potential to improve decision-making and revolutionize care of AIS patients in Hong Kong and globally. Clinicians will be able to utilize our results to provide the best and most cost-effective timing for initiating brace treatment.

DETAILED DESCRIPTION:
Bracing is the mainstay treatment for preventing adolescent idiopathic scoliosis (AIS) progression and the main purpose for treatment is to prevent deformities from reaching the surgical threshold. It has been shown to be effective at reducing curve progression especially in patients with good compliance to treatment. However, bracing should not be used indiscriminately as certain complications have been reported. Bracing too early is safe for curve control but may subject children to prolonged discomfort with the bracing and increased consumption of resources for periodic brace fabrication. Prolonged bracing also reduces spinal mobility, lead to poor body image and self-esteem, and worsen quality of life. Additional risks of osteoporosis and muscular atrophy may also occur. Hence, being able to initiate prompt and appropriate bracing is crucial for achieving optimal curve control and avoiding complications.

Yet, there are still have difficulties identifying patients who may deteriorate. Generally speaking, skeletally immature AIS patients with curves of 20-40 degrees should consider bracing. However, not all of these patients require bracing and some may not need any treatment. More importantly, the resulting curve magnitude on radiographs may not correlate directly with health-related quality of life (HRQOL) measures. As such, the relationship of the Cobb angle prior to initiating brace treatment with long-term HRQOL measures is unknown. The above suggest that there is a significant gap in our knowledge of the optimal timing of brace initiation for managing AIS patients.

In the current setting of rising health-care expenditures, it is also important to assess the "value" of management options and provide the best and cost-effective care for our AIS patients without compromising outcomes or safety. Some clinicians may be more aggressive by bracing children with minor curves while some are content with prescribing braces only when deterioration occurs in moderate curves. In this modern era of healthcare, there is increasing emphasis placed on monitoring and controlling health-care costs to the patient, hospital and insurance companies. Hence, it is an appropriate time to consider the relationship of cost-effectiveness factors and HRQOL measures in designing bracing protocols for AIS patients. With increasing health-care costs, consumption of resources, and the imperative to provide the best healthcare to these children, and focus on a cost-effective delivery of care.

It is thus timely for us to perform this prospective cost-effectiveness comparative study to identify the best indications for initiating brace treatment for AIS patients. Evidence for the best HRQOL outcomes at the lowest cost from both the patient and health-care perspective is necessary to further improve the care for AIS patients. There is potential for the derived model to be applied in other healthcare systems by using a more personalized approach.

For this study, the investigators will utilize mathematical modeling based on factors including initial Cobb angle, maturity status, brace duration, and HRQOL measures to determine the best cost-effective indications for brace treatment. Outcomes will be dependent on the Cobb angle at the end of bracing, HRQOL measures and the overall costs incurred to patients and infrastructure. Our hypothesis is given an AIS patient with significant growth potential, a Cobb angle of 25 degrees is most cost-effective for initiating bracing. On the contrary, bracing for subjects with Cobb angles of 40 degrees or more is not cost-effective regardless of remaining growth.

The main objectives of this study are:

1. To assess the cost-effectiveness of current bracing protocols for AIS.
2. To create a mathematical model that will determine the most cost-effective threshold for initiating brace treatment based on health quality of life measures.

This is a prospective comparative cost-effectiveness analysis between bracing groups. This study will be carried out at the Duchess of Kent Children's Hospital (DKCH). Prospective collection of data from AIS patients including clinical and radiographic information. The investigators will only include AIS patients seen in the first setting with remaining growth potential (Risser 0-2) that may be considered for bracing, and will be prescribed with either underarm (Boston) or Milwaukee bracing. The investigators will collect a minimum of two-year longitudinal data, having at least 5 follow-up data points or clinic visits. It is clinic protocol that all subjects undergo weight, height and arm span measurements, radiographs and doctor assessments at these visits. For this study, HRQOL and utility measurements are vital to its success. Thus, the SRS-22r and EQ-5D-5L questionnaire will be provided at every visit. Three subgroups for analysis between groups. For groups of baseline Cobb angles (20-<35, 35-40, >40 degrees)

Direct and indirect cost will be analyzed. The medical cost (direct costs) for each patient since the first presentation will be obtained. The cost includes the expenses for clinic follow-up, any form of outpatient and inpatient treatment (including physiotherapy, scoliosis specific exercises, bracing) and complications. Unit cost of investigation, treatment and follow-up will be based on the Hospital Authority official charges to non-eligible persons available in the 2013 Hong Kong Government Gazette and updated charges in Hospital Authority website. Brace costs include the number of orthotic visits, per visit consultation cost for the orthotist fabrication of the brace, consumables for use, number of exchanges or modifications, and the thermal sensor for monitoring compliance. In addition to the orthotist, other allied health professionals are also part of the bracing program which further increases the cost. Physiotherapists are involved to maintain body posture and teach/perform scoliosis specific exercises. A clinical psychologist will periodically assess the patient and family to maintain mental health. will be included in the cost analysis. For subjects with failed conservative treatment meaning progression of the curve and no longer indicated for bracing or further bracing will undergo surgical intervention. These subjects are still analyzed but an addition cost item of "surgery" (one lump-sum to cover general cost of implants, hospital length of stay, operating theater cost) will be included. The cost of family members missing work (indirect costs) will also be assessed.

Cost-effectiveness analysis of initiating for bracing will be performed via Markov modelling that will simulate the clinical management of AIS patients since first presentation assuming at age of 11 years (female). Each patient starting at the assumed age 11 will thus follow an annual cycle with a time horizon until 18 years of age. Modelling will be carried out for the AIS patients as a whole, and by the 5 Cobb angle magnitude groups (20-25 degrees, >25-30 degrees, >30-35 degrees, >35-40 degrees, and >40 degrees). For each cycle year, patients initiating bracing may wear the brace until maturity, stop wearing (compliance rate), or switch to surgical approach over the years. Patients with failed bracing will proceed to surgery, and stay with a post-operation health status from operation date to the end. Costs and utility data for AIS patients initiating bracing will be obtained from above prospective study. Clinical model parameters related to compliance rate of bracing, maturity rate of bracing, probability of treatment switch from bracing to surgery will also be identified through a comprehensive review of local and overseas literature as reference. Based on the regression model found, the investigators will estimate the effects of bracing at variable initial curvature and maturity status on direct and indirect costs, SRS-22r domain and total scores, and EQ-5D utility scores. The cost-effectiveness analysis will also recommend a threshold of curvature and maturity combination to indicate when bracing initiated will be the most cost-effective or even cost-saving treatment option for AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with adolescent idiopathic scoliosis and are seen in the first setting with remaining growth potential (Risser 0-2), and are prescribed with either underarm (Boston) or Milwaukee bracing

Exclusion Criteria:

* Patients whose diagnosis is not adolescent idiopathic scoliosis, unable to comply with study follow-up and refused consent for study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a prospective cohort of AIS patients who are newly prescribed with bracing treatment
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cobb angle | up to 3 years
  Cobb angle changes from final visit as compared to baseline
Cost-effectiveness of bracing - direct and indirect costs | up to 3 years
  Costs involve number of clinic follow-up, any form of outpatient and inpatient treatment (including physiotherapy, scoliosis specific exercises, bracing) and complications. Unit cost of investigation, treatment and follow-up. These will be analyzed against the benefits of bracing on clinical parameters, that is, any deterioration of Cobb angle
Change in C7-CSVL | up to 3 years
  Changes in C7-central sacral vertical line with brace follow-up
Change in truncal shift | up to 3 years
  Changes in truncal shift with brace follow-up
Change in sagittal vertical axis | up to 3 years
  Change sagittal vertical axis with brace follow-up
Change in thoracic kyphosis | up to 3 years
  Change in thoracic kyphosis with brace follow-up
Change in lumbar lordosis | up to 3 years
  Change in lumbar lordosis with brace follow-up
Change in rotational profile | up to 3 years
  Change in 3D parameters/apical rotation with brace follow-up

SECONDARY OUTCOMES:
Patient's quality of life - SRS-22r | up to 3 years
  Using the refined Chinese version of the Scoliosis Research Society-22 (SRS-22r) questionnaire scores changes of total score and domain scores (Domains: Activity, Self-image, Pain, Mental Health, Satisfaction with Treatment). The highest score is 5 for total score and each domain score. The higher the score, the better the patient's quality of life is.
  Total
Patient's quality of life - EQ5DY | up to 3 years
  Using the changes of EQ5DY scores (total score and dimension scores: Mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and EQ-visual analogue scale (EQ-VAS)). Each dimension has 5 levels of response and each response will provide one digit to represent it. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. These health states can be converted into a single index value by using the standard EQ-value sets for the local population. For the EQ-VAS, it is a patient's perception of own general health status on a scale from 0 to 100, with higher the score, the better the status.
Brace compliance | up to 3 years
  Thermal sensor objective compliance data

CONTACTS AND LOCATIONS:
Overall Officials: Jason Cheung, MBBS, MS, Principal Investigator — HKU/HA
Locations (2):
- Hong Kong (2):
  - Duchess of Kent Children's Hospital, Hong Kong
  - Jason Pui Yin Cheung, Hong Kong